CLINICAL TRIAL: NCT06614803
Title: Regulatory Effects of Transcutaneous Auricular Vagus Nerve Stimulation Combined with Slow Breathing on Insomnia and Its Impact on Interoceptive Indicators
Brief Title: Study of the Effects of Transcutaneous Auricular Vagus Nerve Stimulation Combined with Slow Breathing on Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xidian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240731
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Insomnia
Keywords: Insomnia; Interoception; Transcutaneous Auricular Vagus Nerve Stimulation; Slow Breathing
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hypoventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- taVNS combined with slow breathing (Active Comparator): For taVNS combined with slow breathing group,after preparing the skin with an alcohol pad, electrodes were attached to the tragus and cymba conchae of the left ear,and under the guidance of the device's video, the participants were instructed to perform six slow and relaxed breaths per minute (0.1Hz), while the built-in parameters of the device delivered stimulation during the 5 seconds of exhalation.The stimulation parameters were set to a burst pulse wave with a frequency of 20Hz, 200μs, and a burst frequency of 2000Hz, 5s ON-5s OFF;stimulation time:20min.
  Interventions: Device: Transcutaneous vagus nerve stimulation combined slow breathing
- taVNS with normal breathing (Active Comparator): For taVNS with normal breathing group,without video guidance on the stimulation device, the participants breathed freely while receiving normal tVNS intervention.Electrodes were attached to the tragus and cymba conchae of the left ear. The stimulation parameters were set to a burst pulse wave with a frequency of 20Hz, 200μs, 5s ON-5s OFF, and a burst frequency of 2000Hz, ;stimulation time:20min.
  Interventions: Device: Transcutaneous vagus nerve stimulation
- slow breathing with sham taVNS (Active Comparator): For slow breathing with sham taVNS group,the participants followed the video instructions to perform slow breathing while wearing the stimulation electrodes, but the device only outputted stimulation for one minute and then stopped.
  Interventions: Device: Transcutaneous vagus nerve stimulation combined slow breathing
- normal breathing with sham taVNS (Sham Comparator): For normal breathing with sham taVNS group,the device were set to output stimulation for only one minute and then stop, and the participants breathed normally
  Interventions: Device: Transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation combined slow breathing — The stimulation parameters were set to a burst pulse wave with a frequency of 20Hz, 200μs,5s ON-5s OFF,and a burst frequency of 2000Hz. Electrodes were attached to the tragus and cymba conchae of the left ear,the screen of the device displays slow breathing guidance video at 0.1Hz, while the device delivered stimulation during the 5 seconds of exhalation.
  Arms: slow breathing with sham taVNS; taVNS combined with slow breathing
Device: Transcutaneous vagus nerve stimulation — Without slow breathing guidance video on the stimulation device,the stimulation parameters were set to a burst pulse wave with a frequency of 20Hz, 200μs,5s ON-5s OFF,and a burst frequency of 2000Hz. Electrodes were attached to the tragus and cymba conchae of the left ear
  Arms: normal breathing with sham taVNS; taVNS with normal breathing

SUMMARY:
The study recruited college students with insomnia disorders and applied transcutaneous auricular vagus nerve stimulation(taVNS) combined with slow breathing. The main aims of the study are: 1) to explore the role of this novel and effective physical therapy technique of taVNS combined with slow breathing in regulating insomnia; 2) to investigate the relationship between the synergistic effect of taVNS and slow breathing on interoceptive indicators and their therapeutic effects.

DETAILED DESCRIPTION:
This study conducted a randomized controlled clinical trial with an intention to enroll 80 insomnia participants. Participants were randomly assigned in a 1:1:1:1 ratio to four groups:1）taVNS combined with slow breathing group；2）taVNS with normal breathing group；3）slow breathing with sham taVNS group；4）normal breathing with sham taVNS group.The study included a one-week baseline period, a two-week treatment period, and a two-week follow-up period. During the 2-week treatment period, 20 minutes of continuous treatment was performed every evening. The stimulation parameters were set to 20Hz, 200μs, 5s ON-5s OFF and a burst frequency of 2000Hz. For taVNS combined with slow breathing group,after preparing the skin, electrodes were attached to the tragus and cymba conchae of the left ear,and under the guidance of the device's video, the participants were instructed to perform six slow and relaxed breaths per minute (0.1Hz), while the device delivered stimulation during the 5 seconds of exhalation.For taVNS with normal breathing group,without video guidance on the device, the participants breathed freely while receiving normal taVNS intervention.For slow breathing with sham taVNS group,the participants followed the video instructions to perform slow breathing while wearing the stimulation electrodes, but the device only outputted stimulation for one minute.For normal breathing with sham taVNS group,the device outputted stimulation for only one minute, and the participants breathed normally. EEG and ECG data were collected before and after the 2-week treatment, and scale data were collected before and after the treatment as well as at the end of follow-up. Sleep diaries were recorded throughout the 5-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years;
2. Meet the definition of insomnia in the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V)；
3. Has not received any psychotropic drug treatment；
4. PSQI(Pittsburgh Sleep Quality Index) score>7；
5. ISI(Insomnia Severity Index) score≥11；
6. Signed informed consent form;
7. Ability and willingness to comply with the study requirements.

Exclusion Criteria:

1. There are learning or working hours that affect the circadian rhythm;
2. There is abuse of alcohol, nicotine, or other substances;
3. Pregnancy, breastfeeding, or plans to become pregnant;
4. Damage or allergy to the selected stimulation site;
5. Clinically diagnosed mental disorders and other medical conditions;
6. Currently taking stimulant, hormone, or other medications that may cause insomnia and are not suitable for discontinuation.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Sleep diary indicators after two weeks of treatment | Sleep diaries were collected daily for five weeks, but changes in sleep diary data were assessed after one week baseline, two weeks of treatment, and two weeks of follow-up.
  Sleep latency, sleep efficiency, wake time after sleep onset, number of wake times after sleep onset, and total sleep time were used as the primary outcome measure in the sleep diary.

SECONDARY OUTCOMES:
Changes in heart rate variability | Heart rate variability will be assessed twice within five weeks:at baseline,and after two weeks of treatment.
  Heart rate variability(HRV) were analyzed to evaluate the mean peak interval (MeanRR) of the RR and three commonly used measures of autonomic nervous function: the root mean square sum of the difference between adjacent normal heartbeat intervals (RMSSD), the percentage of adjacent NN differences greater than 50ms in the total number of sinus heart beats (PNN 50%), and high frequency power (aHF).
Changes in heartbeat evoked potential | Heartbeat evoked potential will be assessed twice within five weeks:at baseline,and after two weeks of treatment.
  Heartbeat evoked potential(HEP) is the electrical activity of the brain at a specific moment in the heart cycle, which is synchronized with the R wave of the heart's electrical signals and can be measured by recording the electrical activity of the brain at a specific point in time within the heartbeat cycle. HEP represents an electrophysiological marker of cortical processing of incoming cardiovascular information.
Changes in ISI scores | ISI will be assessed three times within five weeks: at baseline, after two weeks of treatment, and two weeks of follow-up.
  The Insomnia Severity Index (ISI) is utilized to assess the severity of insomnia and its impact on physical health, daily function, and quality of life. This scale includes seven items, with a total scoring range from 0 to 28. Higher scores denote more severe insomnia. The change in ISI score will be determined by subtracting the baseline score from the score at each subsequent time point.
Changes in PSQI scores | PSQI will be assessed three times within five weeks: at baseline, after two weeks of treatment, and two weeks of follow-up.
  The Pittsburgh Sleep Quality Index(PSQI) assessed the sleep quality of the participants in the last 1 month, which was composed of 19 self-rated items and 5 other rated items, in which the 19th self-rated items and 5 other rated items did not participate in the score. The 18 self-rated entries that participate in the scoring can be combined into seven sections. They were: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, hypnotic drug use and daytime dysfunction. Each part is scored from 0 to 3, and the cumulative score of each part is divided into PSQI total score, ranging from 0 to 21, and the higher the score, the worse the sleep quality
Change in PHQ-9 scores | PHQ-9 will be assessed three times within five weeks: at baseline, after two weeks of treatment, and two weeks of follow-up.
  The Patient Health Questionnaire-9 (PHQ-9) encompasses nine items, each representing a different facet of depressive symptoms. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms. The change in PHQ-9 score will be determined by subtracting the baseline score from the score at each subsequent time point.
Change in GAD-7 scores | GAD-7 will be assessed three times within five weeks: at baseline, after two weeks of treatment, and two weeks of follow-up.
  The Generalized Anxiety Disorder Scale (GAD-7) is used to assess the emotional state of patients. The Generalized Anxiety Disorder Scale (GAD-7) comprises seven items, with a total possible score ranging from 0 to 21. An elevated score suggests a more pronounced level of anxiety. The change in GAD-7 score will be determined by subtracting the baseline score from the score at each subsequent time point.
Change in FFS scores | FFS will be assessed three times within five weeks: at baseline, after two weeks of treatment, and two weeks of follow-up.
  The Flinders Fatigue Scale(FFS) consists of seven entries that measure various fatigue characteristics (e.g., frequency, severity) experienced during the past two weeks. Six items were presented in Likert form, with responses ranging from 0(not at all) to 4(very serious). The total score is calculated by the sum of all the items. The total score of the scale ranges from 0 to 31 points, and the higher the score, the more serious the fatigue degree of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Wei, Phd, Principal Investigator — Xidian University
Locations (1):
- Xidian University, Xi'an, Shaanxi, China